CLINICAL TRIAL: NCT00702923
Title: Phase I Dose Escalation Trial of CP-675,206 (Tremelimumab, Anti-CTLA-4 Monoclonal Antibody) in Combination With Short Term Androgen Deprivation in Patients With Stage D0 Prostate Cancer
Brief Title: CP-675,206 in Combination With Short Term Androgen Deprivation in Patients With Stage D0 Prostate Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Enrollment was halted prematurely due to slow accrual.
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CO07808; CO07808; H-2008-0086 (Other: Institutional Review Board); NCI-2011-00713 (Registry Identifier: NCI Trial ID); A534260 (Other: UW Madison); SMPH/MEDICINE/MEDICINE*H (Other: UW Madison)
Record Dates: First submitted 2008-06-18; First posted 2008-06-20 (Estimated); Results first posted 2014-05-07 (Estimated); Last update posted 2019-11-21 (Actual); Status verified 2014-04

CONDITIONS: Prostate Cancer
Keywords: Stage D0 Prostate Cancer; Rising PSA; Casodex; Tremelimumab
MeSH Terms: conditions — Prostatic Neoplasms | interventions — bicalutamide; tremelimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Bicalutamide 150mg orally days 1-28 followed by CP-675,206 IV on day 29. Cycle is repeated once at month 3
  Interventions: Drug: Bicalutamide and CP-675,206 (Tremelimumab); Drug: Bicalutamide, CP-675,206 (tremelimumab); Drug: Bicalutamide, CP-675,206

INTERVENTIONS:
Drug: Bicalutamide and CP-675,206 (Tremelimumab) — Dose level -1 :
  Bicalutamide 150 mg p.o. q.d. day 1-28 CP-675,206 3 mg/kg I.V. over 1 hour, day 29 Cycle repeated once at month 3 (beginning day 85 +/- 7)
  Other Names: Casodex; Tremelimumab
Drug: Bicalutamide, CP-675,206 (tremelimumab) — Dose level 1:
  Bicalutamide 150 mg p.o. q.d. day 1-28 CP-675,206 6 mg/kg I.V. over 1 hour, day 29 Cycle repeated once at month 3 (beginning day 85 +/- 7)
  Other Names: Casodex; Tremelimumab
Drug: Bicalutamide, CP-675,206 (Tremelimumab) — Dose level 2:
  Bicalutamide 150 mg p.o. q.d. day 1-28 CP-675,206 10 mg/kg I.V. over 1 hour, day 29 Cycle repeated once at month 3 (beginning day 85 +/- 7)
  Other Names: Casodex; Tremelimumab
Drug: Bicalutamide, CP-675,206 (Tremelimumab) — Dose level 3:
  Bicalutamide 150 mg p.o. q.d. day 1-28 CP-675,206 15 mg/kg I.V. over 1 hour, day 29 Cycle repeated once at month 3 (beginning day 85 +/- 7)
  Other Names: Casodex; Tremelimumab
Drug: Bicalutamide, CP-675,206 — Final Dose Level:
  Bicalutamide 150 mg p.o. q.d. day 1-28, day 85-112
  At month 9, if evidence of PSA progression:
  Bicalutamide 150 mg p.o. q.d. day 1-28 CP-675,206 (MTD dose) I.V. over 1 hour, day 29
  Other Names: Casodex; Tremelimumab

SUMMARY:
The current protocol will evaluate the safety of combining treatment with bicalutamide(Casodex) and CP-675,206 (anti-CTLA-4 monoclonal antibody) in patients with PSA-recurrent non-metastatic (stage D0) prostate cancer. This is a dose escalation study with safety the primary endpoint. Secondary endpoints will be to determine whether prostate associated immune responses are seen, and whether treatment is associated with an increase in PSA doubling time and PSA recurrence at one year, as markers of clinical activity. Cohorts of six patients will be treated in each dose level. The investigators hypothesize that short-term androgen deprivation therapy will elicit prostate cancer-associated T-cell mediated tissue destruction that can be augmented with a monoclonal antibody blocking CTLA-4, and that this will have therapeutic benefit in patients with recurrent prostate cancer.

DETAILED DESCRIPTION:
This is an open label, single-center Phase I study. All subjects will receive bicalutamide 150mg orally days 1-28. Subjects will receive CP-675,206 IV over one hour on day 29. Doses will range from 6 mg/kg to 15 mg/kg. This cycle will be repeated once at month 3. Once the maximum tolerated dose has been determined, up to 6 additional subjects will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age & histologic diagnosis of adenocarcinoma of the prostate
* Completed surgery or radiation at least 8 weeks prior to entry with removal of all visible disease
* Clinical Stage D0 prostate cancer with rising PSA and PSA >2ng/ml.
* ECOG performance of <2
* Normal hematologic, renal and liver function

Exclusion Criteria:

* Cannot have evidence of immunosuppression or have been treated with immunosuppressive therapy.
* No prior treatment with an LHRH agonist or nonsteroidal antiandrogen such as casodex or flutamide
* No evidence for metastatic disease per bone scan or CT scan of the abdomen and pelvis
* No prior treatment with anti-CTLA 4 monoclonal antibody
* No history of known autoimmune disorder or HIV, hepatitis B or hepatitis C
* No known brain metastases
* No history of inflammatory bowel conditions including diverticulitis, ulcerative colitis, etc.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2008-07; Primary Completion 2011-09 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas McNeel, MD, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Paul P. Carbone Comprehensive Cancer Center, Madison, Wisconsin, United States

REFERENCES:
- See also: University of Wisconsin Carbone Cancer Center — https://cancer.wisc.edu/

RESULTS

PARTICIPANT FLOW:
Groups:
- CP-675,206 in Combination With Short Term Androgen Deprivation: Bicalutamide 150mg orally days 1-28 followed by CP-675,206 IV on day 29. Cycle is repeated once at month 3
Period: Overall Study
Arm/Group | CP-675,206 in Combination With Short Term Androgen Deprivation
Started | 12
Completed | 11
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | CP-675,206 in Combination With Short Term Androgen Deprivation
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.7 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 12
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants Who Developed Cancer Antigen-specific Immune Responses
Time Frame: Up to 12 months after treatment with study agent
Measure: Number; unit: participants
Groups:
- CP-675,206 3mg/kg: Dose level -1: Bicalutamide 150mg orally once a day on days 1-28 and CP-675,206 3mg/kg intravenously over 1 hour on day 29. The treatment is repeated at month 3 (beginning day 85).
- CP-675,206 6mg/kg: Dose level 1: Bicalutamide 150mg orally once a day on days 1-28 and CP-675,206 6mg/kg intravenously over 1 hour on day 29. The treatment is repeated at month 3 (beginning day 85).
Arm/Group | CP-675,206 3mg/kg | CP-675,206 6mg/kg
Number analyzed (Participants) | 6 | 5
participants
  one or more prostate-associated antigens | 6 | 5
  antibodies specific for PSA | 2 | 1

2. Secondary Outcome: The Number of Participants With an Increase in PSA Doubling Time
Time Frame: Up to 18 months after last dose of study agent
Measure: Number; unit: participants
Arm/Group | CP-675,206 3mg/kg | CP-675,206 6mg/kg
Number analyzed (Participants) | 6 | 5
participants
  immediate post-treatment period (6-12 months) | 0 | 0
  12-18 months after treatment | 2 | 1

3. Secondary Outcome: Number of Participants With PSA Recurrence.
Description: PSA recurrence is defined as a minimum PSA value of greater or equal to 1.0ng/ml occurring within one year after the last treatment with CP-675,206, with a confirmatory PSA blood teat performed at least 2 weeks later.
Time Frame: one year
Measure: Number; unit: participants
Arm/Group | CP-675,206 3mg/kg | CP-675,206 6mg/kg
Number analyzed (Participants) | 6 | 5
participants | 6 | 5

ADVERSE EVENTS:
Arm/Group | CP-675,206 in Combination With Short Term Androgen Deprivation
Serious Adverse Events (participants affected / at risk) | 1/12
Other Adverse Events (participants affected / at risk) | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CP-675,206 in Combination With Short Term Androgen Deprivation (N=12)
Autoimmune Reaction (Immune system disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CP-675,206 in Combination With Short Term Androgen Deprivation (N=12)
Constipation (Gastrointestinal disorders) | 2 (2)
Allergic Rhinitis (Immune system disorders) | 2 (2)
Autoimmune Reaction (Immune system disorders) | 1 (1)
Hypertension (Cardiac disorders) | 1 (1)
Hypotension (Cardiac disorders) | 1 (1)
Fatigue (General disorders) | 7 (11)
Fever (General disorders) | 1 (1)
Rigors/chills (General disorders) | 2 (2)
Weight Loss (General disorders) | 1 (1)
Dermatology/Skin-Other (Skin and subcutaneous tissue disorders) | 3 (4)
Dry Skin (Skin and subcutaneous tissue disorders) | 1 (1)
Hair Loss/Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 4 (5)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 3 (3)
Acne/acneiform (Skin and subcutaneous tissue disorders) | 4 (6)
Hot flashes/flushes (Endocrine disorders) | 4 (6)
Anorexia (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 3 (9)
Distension/bloating, abdominal (Gastrointestinal disorders) | 2 (3)
Gastrointestinal--Other (Gastrointestinal disorders) | 1 (1)
Incontinence, anal (Gastrointestinal disorders) | 1 (1)
Mucositis/sttomatitis (clinical exam)--Oral Cavity (Gastrointestinal disorders) | 2 (3)
Mucositis/stomatitis (functional/symptomatic) --Anus (Gastrointestinal disorders) | 1 (1)
Mucositis/stomatits (functional/symptomatic)--Oral Cavity (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (5)
Hemorrhage, GU--Bladder (Renal and urinary disorders) | 1 (1)
Hemorrhage, Gu--Urinary NOS (Renal and urinary disorders) | 2 (2)
Hemorrhage/bleeding--Other (Renal and urinary disorders) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils--Sinus (Infections and infestations) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils--Skin (Infections and infestations) | 1 (1)
Edema: limb (Blood and lymphatic system disorders) | 2 (2)
Amylase (Investigations) | 1 (2)
Fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness, generalized or specific area--Extremity-lower (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Mood alteration--Agitation (Nervous system disorders) | 1 (1)
Mood alteration--Anxiety (Nervous system disorders) | 1 (1)
Mood alteration--Depression (Nervous system disorders) | 2 (4)
Neurology--Other (Nervous system disorders) | 1 (1)
Dry eye syndrome (Eye disorders) | 1 (1)
Ocular/Visual--Other (Eye disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Voice changes/dysarthiria (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Renal/Genitourinary--Other (Renal and urinary disorders) | 1 (2)
Urinary frequency/urgency (Renal and urinary disorders) | 2 (2)
Urinary retention (Renal and urinary disorders) | 2 (3)
Gynecomastia (Reproductive system and breast disorders) | 4 (4)
Pain--Abdomen NOS (Gastrointestinal disorders) | 4 (6)
Pain - Breast (Reproductive system and breast disorders) | 3 (3)
Pain - Head/headache (Nervous system disorders) | 1 (1)
Pain - Joint (Musculoskeletal and connective tissue disorders) | 1 (1)
flu-like syndrome (General disorders) | 1 (1)
Pain - neck (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes